CLINICAL TRIAL: NCT02409134
Title: Cognitive Function and Patient-Reported Psychological and Functional/Quality of Life Outcomes Investigation in Patients Taking Vorinostat for Graft-versus-Host Disease Prophylaxis
Brief Title: Cognitive Function and Patient-Reported Quality of Life Outcomes Investigation in Patients Taking Vorinostat
Status: Completed | Type: Observational
Sponsor: Sung Choi, M.D. (Other)
Responsible Party: Sponsor-Investigator, Sung Choi, M.D., Assistant Professor, University of Michigan Rogel Cancer Center
Organization: University of Michigan Rogel Cancer Center (Other)
Other Study IDs: UMCC 2015.020; HUM00096406 (Other: University of Michigan Cancer Center)
Record Dates: First submitted 2015-03-23; First posted 2015-04-06 (Estimated); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: Quality of Life; Graft-vs-Host Disease
Keywords: Bone Marrow Transplantation; Hematologic Malignancies; Adults; Cognition
MeSH Terms: conditions — Graft vs Host Disease; Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Psychological well-being and cognitive function will be measured in patients enrolled on the primary study, NCT01790568, a phase 2 trial of vorinostat plus tacrolimus and methotrexate to prevent graft versus host disease following unrelated donor hematopoietic stem cell transplantation. Validated questionnaires will be administered to assess patients' level of depression, anxiety, quality of life, perceived cognitive functioning, and sleep quality. Cognitive testing will include reliable and valid measures of processing speed, attention, executive function, episodic memory, and visual learning and memory. The purpose of this study is to determine whether these measures are feasible to administer in patients before and at early time points after bone marrow transplantation .

ELIGIBILITY:
Inclusion Criteria:

* Patients must be enrolled on the parent study (NCT01790568; A phase 2 clinical trial of vorinostat plus tacrolimus and methotrexate to prevent graft versus host disease following unrelated donor hematopoietic stem cell transplantation)
* Must speak, read and understand English

Exclusion Criteria:

* Documented evidence of cognitive impairment prior to enrollment on this study (diagnosis of dementia, mild cognitive impairment, or other neurological illnesses that impact cognition).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients enrolled on the primary study NCT01790568. Eligible patients who choose not to participate in this add-on study will not be excluded from participating in NCT01790568.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2015-04; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Feasibility, as measured by completion of cognitive testing and validated questionnaires at all time points by 50% of newly-accrued patients. | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan Health System, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Hoodin F, LaLonde L, Errickson J, Votruba K, Kentor R, Gatza E, Reddy P, Choi SW. Cognitive Function and Quality of Life in Vorinostat-Treated Patients after Matched Unrelated Donor Myeloablative Conditioning Hematopoietic Cell Transplantation. Biol Blood Marrow Transplant. 2019 Feb;25(2):343-353. doi: 10.1016/j.bbmt.2018.09.015. Epub 2018 Sep 20. PMID 30244099